CLINICAL TRIAL: NCT07322653
Title: Prospective, Open-Label, Multicenter Study to Characterise the Effects of Co-administration of MediDrink Platinum+ Formula Containing Novel Protein Blend SPR-01 and Fava Bean Protein Hydrolysate on Fitness in an Aged Population
Brief Title: The Effects of MediDrink Platinum+ and Fava Bean Protein Hydrolysate on Fitness in an Aged Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Collaborators: Medifood Hungary Innovation Kft (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SPR-K-2024-01; GINOP PLUSZ 2.1.1-21-102200048 (Other Grant/Funding Number: GINOP PLUSZ)
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia in Elderly; Malnourished; Protein Supplementation; Muscle Mass; Physical Function; Strength
Keywords: Sarcopenia; Peptide Therapeutics; PeptiStrong; MediDrink Platinum; Malnourished Elderly; Physical functioning; MediDrink Platinum+; Clinical Nurtition; Nutritional status
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Intervention Model Description: All participants begin on the base formula MediDrink Platinum before splitting into one of two arms, the version containing novel protein blend SPR-01, MediDrink Platinum+, or MediDrink Platinum+ and 2.4g of PeptiStrong supplement
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MediDrink Platinum+ (Active Comparator): Base formula containing novel protein blend SPR-01 (Dosed appropriate to nutritional status with a minimum of 1200kcal/day as 600ml)
  Interventions: Other: MediDrink Platinum+
- MediDrink Platinum+ and PeptiStrong (Experimental): Base formula containing novel protein blend SPR-01 (Dosed appropriate to nutritional status with a minimum of 1200kcal/day as 600ml) and 2.4g/day PeptiStrong
  Interventions: Other: MediDrink Platinum+ and PeptiStrong

INTERVENTIONS:
Other: MediDrink Platinum+ — MediDrink Platinum+ containing novel protein blend SPR-01
  Other Names: Clinical Nutrition
  Arms: MediDrink Platinum+
Other: MediDrink Platinum+ and PeptiStrong — MediDrink Platinum+ containing novel protein blend SPR-01 and PeptiStrong, fava bean protein hydrolysate
  Other Names: Clinical Nutrition
  Arms: MediDrink Platinum+ and PeptiStrong

SUMMARY:
Examining the effects of MediDrink Platinum+ containing novel protein blend SRP-01 alone or when combined with PeptiStrong on clinical responses in elderly adults with sarcopenia

DETAILED DESCRIPTION:
The primary aim of this multicentre randomised active control group study , is to characterise the effect of MediDrink Platinum+ containing a novel protein blend SPR-01, alone and in combination with PeptiStrong on general fitness measured via the Barthel index in malnourished sarcopenic, adults, aged 60 and above. The trial will incorporate a "Y" design whereby all 75 participants begin on the base formula (MediDrink Platinum) for 2 weeks before being randomised into the SPR-01 alone (n=37, dose calculated per individual but at least 1200 kcal/day) or SP1-01 and PeptStrong (n=38, dose calculated per individual but at least 1200 kcal per day and 2.4g/day, respectively) supplementation arms for 10 weeks.

Other clinical endpoints measured as secondary endpoints will include hand grip strength, physical functioning via time up&go test and changes in fat-free body mass.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* BMI ≤ 25 kg/m²
* Malnourished (mini nutritional assessment MNA <11
* Sarcopenic: SARC-F score ≥ 4
* Capable or oral feeding either alone or assisted
* Ambulatory (WHO PS/ECOG 0-3)
* Ability to complete questionnaires and self assess health status
* Ability to provide consent

Exclusion Criteria:

* Patient cannot eat orally
* Acute Infection
* Proven Intestinal obstruction
* Co-morbidities requiring a special diet (diabetes, kidney disease etc.)
* Liver dysfunction
* Acute or chronic renal failure
* Uncontrollable nausea or vomiting
* Use of megestrol acetate or metabolic steroids
* Dietary supplement use in the last 3 months
* Known intolerance or allergy to the investigational products
* Participation in any clinical trial within the last 3 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
General well-being via Barthel Index | Whole group Week 0 to Week 2. Investigational arms Week 2 to Week 12
  Time to 5 point change in Barthel Index compared from baseline (visit 0) to week 2 in the whole patient population versus week 2 to week 12 in the two investigational groups; MediDrink Platinum+ and MediDrink Platinum+ with PeptiStrong.
  The Barthel scale measures the ability to perform basic activities of daily living using 10 variables describing mobility. A higher value is associated with a higher likelihood of independence

SECONDARY OUTCOMES:
Hand Grip Strength via Dynamometer | Whole group Week 0 to Week 2. Investigational arms Week 2 to Week 12
  Change in hand grip strength compared from baseline (Visit 0) to week 2 in the whole patient population versus week 2 to week 12 in the two investigational groups; MediDrink Platinum+ and MediDrink Platinum+ with PeptiStrong.
Fat-free body mass via bioelectrical impedance analysis | Whole group Week 0 to Week 2. Investigational arms Week 2 to Week 12
  Change in fat-free body mass compared from baseline (visit 0) to week 2 in the whole patient population versus week 2 to week 12 in the two study groups; MediDrink Platinum+ and MediDrink Platinum+ with PeptiStrong.
Functional performance via time up & go test | Whole group Week 0 to Week 2. Investigational arms Week 2 to Week 12
  Change in time to up & go compared from baseline (visit 0) to week 2 in the whole patient population versus week 2 to week 12 in the two study groups; MediDrink Platinum+ and MediDrink Platinum+ with PeptiStrong.

OTHER OUTCOMES:
General well-being via Barthel Index (Active control Vs experimental) | Week 2 to Week 12
  Time to 5 point change in Barthel Index compared from week 2 to week 12 in the two investigational groups; MediDrink Platinum+ and MediDrink Platinum+ with PeptiStrong.
  The Barthel scale measures the ability to perform basic activities of daily living using 10 variables describing mobility. A higher value is associated with a higher likelihood of independence
Hand Grip Strength via Dynamometer ( Active control Vs experimental) | Week 2 to Week 12
  Change in hand grip strength compared from week 2 to week 12 in the two investigational groups; MediDrink Platinum+ and MediDrink Platinum+ with PeptiStrong.
Fat-free body mass via bioelectrical impedance analysis | Week 2 to Week 12
  Change in Fat-free body mass compared from week 2 to week 12 in the two study groups; MediDrink Platinum+ and MediDrink Platinum+ with PeptiStrong.
Functional performance via time up & go test (Active control Vs experimental) | Week 2 to Week 12
  Change in time to up & go compared from week 2 to week 12 in the two study groups; MediDrink Platinum+ and MediDrink Platinum+ with PeptiStrong.

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - Országos Korányi Pulmonológiai Intézet, Budapest
  - Sóstói Szivárvány Idősek Otthona, Nyíregyháza

IPD SHARING:
Plan to Share IPD: No